CLINICAL TRIAL: NCT05521451
Title: Longterm Outcome and Predictors for Recurrence After Medical and Interventional Treatment of Arrhythmias At the University Heart Center Hamburg
Brief Title: Clinical Cohort Study - TRUST
Acronym: TRUST
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: CCS_TRUST
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Ventricular Tachycardia; Atrial Tachycardia; Arrhythmogenic Right Ventricular Dysplasia; Long QT Syndrome; Brugada Syndrome; Supraventricular Tachycardia; Catecholaminergic Polymorphic Ventricular Tachycardia; Torsades De Pointes; Atrial Cardiomyopathy
Keywords: Catheter Ablation; Biomarkers; Cardiac Arrhythmia; eHealth; Digital Cardiology; Echocardiography; Atrial Cardiomyopathy
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Tachycardia, Ventricular; Arrhythmogenic Right Ventricular Dysplasia; Long QT Syndrome; Brugada Syndrome; Tachycardia, Supraventricular; Polymorphic Catecholaminergic Ventricular Tachycardia; Torsades de Pointes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood sampling at baseline: Whole blood, serum, cellular RNA Collection of tissue samples excised in clinical routine (e. g. left atrial appendages after surgical closure)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The "Long-term Outcome and Predictors for Recurrence after Medical and Interventional Treatment of Arrhythmias at the University Heart Center Hamburg" (TRUST) study is an investor-initiated, single-center, prospective clinical cohort study including patients treated with cardiac arrhythmias or at high risk for cardiac arrhythmias. The design enables prospective, low-threshold, near complete inclusion of patients with arrhythmias treated at the UHZ. Collection of routine follow-up data, detailed procedural information and systematic biobanking will enable precise and robust phenotyping.

DETAILED DESCRIPTION:
Arrhythmias such as atrial fibrillation, ventricular tachycardia, and sudden death remain major causes of morbidity and mortality. Their prevalence increases in our ageing populations. Modern therapy of these conditions, using a combination of drugs, devices, and interventions, can reduce the disease burden associated with cardiac arrhythmias. This prospective cohort study will collect detailed clinical, procedural, and outcome information in a large cohort of patients with arrhythmias seen in a tertiary care center. Clinical phenotyping will be enhanced by biosampling and analysis of circulating biomolecules. Digital capture of clinical information and of follow-up data is planned.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrhythmia, including congenital cardiac arrhythmia diagnosed at baseline or high risk for cardiac arrhythmia
* Age ≥ 18 years
* Written informed consent
* Ability to provide written informed consent in accordance with Good Clinical Practice and local legislation

Exclusion Criteria:

* Insufficient knowledge of the German language to understand study documents and interview without translation
* Physical or psychological incapability to cooperate in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in the Department of Cardiology of the University Heart and Vascular Center Hamburg suffering from cardiac arrhythmias, including congenital cardiac arrhythmias, or being at high risk for cardiac arrhythmias.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to a composite of cardiovascular mortality, stroke, acute coronary syndrome and heart failure hospitalization | Follow-up 5 years after inclusion
  The main primary outcome measures the time until any of death from cardiovascular cause, stroke or TIA or a hospitalization due to heart failure or acute coronary syndrome occurs for the first time after inclusion. The outcome is measured via telephone and / or in-person follow-up, acquisition of all relevant medical records between inclusion and follow-up timepoint and a questionnaire sent to the patient. The follow-up can be completed fully electronically according to patient's wish.
New onset of cardiac arrhythmias, documented in clinical care and during systematic rhythm monitoring using digital devices. | Follow-up 5 years after inclusion
  The outcome is measured via remote follow-up using consumer-electronics based remote rhythm monitoring technologies. Additionally, onset of new cardiac arrhythmias is assessed from medical records collected between follow-up timepoint and inclusion as well as questionnaires and a telephone call with the patient.

SECONDARY OUTCOMES:
Time to recurrence of the clinical arrhythmia | Follow-up 5 years after inclusion
  The outcome is measured via remote follow-up using consumer-electronics based remote rhythm monitoring technologies. Additionally, onset of new cardiac arrhythmias is assessed from medical records collected between follow-up timepoint and inclusion as well as questionnaires and a telephone call with the patient.
New onset of heart failure | Follow-up 5 years after inclusion
  This endpoint is defined as a new diagnosis of heart failure with (milly) reduced or preserved ejection fraction according to ESC guidelines. The patients medical record will be reassessed at the end of follow-up.
All-cause mortality (Safety Outcome) | Follow-up 5 years after inclusion
  This endpoint is assessed during the telephone call during remote follow-up and - if not applicable - via consultation of the death registry.
Patient reported quality of life (QOL) | Follow-up 5 years after inclusion
  As assessed via AF Effect on QualiTy of life survey at the timepoint of follow-up.
Health care utilisation | Follow-up 5 years after inclusion
  Health care utilisation after inclusion is assessed during the telephone call of the remote follow-up as well as via acquisition of all medical records between follow-up timepoint and inclusion.
Complications of rhythm control therapy (Safety Outcome) | Follow-up 5 years after inclusion
  This endpoint is assessed during the telephone call of the remote follow-up as well as via acquisition of all medical records between follow-up timepoint and inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Paulus Kirchhof, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Andreas Metzner, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Andreas Rillig, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, University Heart and Vascular Center, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] My I, Moser F, Loeck FW, Obergassel J, Rottner L, Lemoine MD, Kirchhof P, Steven D, Sultan A, Willems S, Meyer C, Reissmann B, Rillig A, Metzner A, Ouyang F. Long-term outcome of catheter ablation of left fascicular ventricular arrhythmias. J Interv Card Electrophysiol. 2026 Jan;69(1):35-41. doi: 10.1007/s10840-025-02116-6. Epub 2025 Aug 14. PMID 40810874
- [Derived] Wenzel JP, Lemoine MD, Rottner L, My I, Moser F, Obergassel J, Nies M, Riess J, Ismaili D, Nikorowitsch J, Ouyang F, Kirchhof P, Rillig A, Metzner A, Reissmann B. Nonthermal Point-by-Point Pulmonary Vein Isolation Using a Novel Pulsed Field Ablation System. Circ Arrhythm Electrophysiol. 2023 Sep;16(9):e012093. doi: 10.1161/CIRCEP.123.012093. Epub 2023 Aug 28. No abstract available. PMID 37638409
- See also: Related Info — https://www.uke.de/kliniken-institute/kliniken/kardiologie/ueber-die-klinik/bereich-rhythmologie/index.html
- See also: Related Info — https://www.uke.de/landingpage/uccs/working-groups/working-group-fabritz/index.html